CLINICAL TRIAL: NCT00287495
Title: Phase I and Pharmacokinetic Study of BAY 43-9006 (Sorafenib) in Patients With Kaposi's Sarcoma
Brief Title: BAY 43-9006 (Sorafenib) to Treat Patients With Kaposi's Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060083; 06-C-0083; NCT00304122 (obsolete NCT alias)
Record Dates: First submitted 2006-02-04; First posted 2006-02-06 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2017-10-18

CONDITIONS: Kaposi's Sarcoma; HHV-8; KSHV
Keywords: AIDS; HIV; Antiangiogenesis; VEGF; AIDS Malignancy; Kaposi Sarcoma; KS
MeSH Terms: conditions — Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome | interventions — Sorafenib

ARMS (2):
- A (Experimental): Patients with AIDS-KS receiving ritonavir will be given 200 mg BAY 43-9006 once daily with dose escalation up to 400 mg twice daily
  Interventions: Drug: BAY 43-9006
- B (Experimental): Patients with AIDS-KS not receiving ritonavir will be given 200 mg BAY 43-9006 once daily with dose escalation up to 400 mg twice daily
  Interventions: Drug: BAY 43-9006

INTERVENTIONS:
Drug: BAY 43-9006 — BAY 43-9006 200 mg once daily with dose escalation up to 400 mg twice daily

SUMMARY:
Background:

* Kaposi's sarcoma (KS) is a disease in which cancer cells are found in the tissues under the skin or mucous membranes that line the mouth, nose, and anus. KS causes red or purple patches (lesions) on the skin or mucous membranes and spreads to other organs in the body, such as the lungs, liver, or intestinal tract.
* BAY 43-9006 inhibits the activity of several proteins or protein receptors in cells that are thought to be important to the progression of KS. Blocking these mechanisms may cause KS to get better.

Objectives:

* To learn about the toxicity and blood levels of BAY 43-9006 in people with KS who are and are not taking the anti-retroviral drug ritonavir.
* To look for evidence of a beneficial treatment effect of BAY 43-9006

Eligibility:

* Adults with confirmed KS, both HIV-positive and HIV-negative.
* Patients must have either 1) at least five measurable KS lesions with no previous local therapy, or 2) other measurable non-skin disease that permits evaluation of a response to treatment.

Design:

* Patients are randomly assigned to a specific dose of BAY 43-9006. They take the drug by mouth either once or twice daily, depending on their dose group, for up to 54 weeks.
* Drug blood levels are determined after patients have been taking BAY 43-9006 for 1 to 2 weeks by blood collections immediately before the dose and at 1, 2, 4, 8, 12, 16 and 24 hours after the dose.
* Patients are evaluated every 3 weeks with review of a medication diary, interview about drug side effects, physical examination, and assessment of KS lesions.
* KS lesions are photographed on entering the study and at other time points during the study.
* CD4 cell counts and HIV viral load are tested every 12 weeks.
* Biopsies are done at the start of the study, on day 15, and if it appears that all of the lesions have resolved.
* Other procedures, such as CT or MRI scans, may be done if medically indicated.

DETAILED DESCRIPTION:
BACKGROUND: This study is designed to test the toxicity and pharmacokinetics of different doses of BAY 43-9006 (Sorafenib) in patients with Kaposi s sarcoma (KS). It will also assess, in a preliminary manner, the activity of BAY 43-9006 in this disease and its effect on biological markers. BAY 43-9006 is a potent inhibitor of wild-type and mutant c-Raf kinase isoforms. In addition, this agent also inhibits p38, c-kit, vascular endothelial growth factor receptor 2(VEGFR2), VEGF-R3, and platelet derived growth factor receptor beta (PDGFR-B). There is evidence that several of these receptors, and especially VEGF-R2, VEGF-R3, and PDGF-RB, are important in KS pathogenesis. The principle tumor cells of KS lesions are spindle cells, which are derived from endothelial cells. Spindle cells proliferate in response to VEGF, VEGF-C (a ligand for VEGF-R3), and PDGF, and the stimulation of spindle cells by these factors appears to be an important component in the pathogenesis of KS. There is also evidence that c-kit is important in KS. Because BAY 43-9006 can inhibit the function of these receptors and c-kit, it may have specific activity against this tumor. BAY 43-9006 is metabolized at least in part by CYP 3A4, and ritonavir, an HIV protease inhibitor commonly used in AIDS patients, is an inhibitor of CYP 3A4. Also, AIDS patients are often quite sensitive to drug toxicities. Thus, patients with AIDS-KS on ritonavir may be particularly sensitive to BAY 43-9006.

OBJECTIVES: To assess the toxicity profile and pharmacokinetics of BAY 43-9006 at oral dose regimens of 200 mg once daily, 200mg twice daily, or 400 mg twice daily, up to the toxic dose, in patients with HIV-associated Kaposi s sarcoma (KS) who are receiving ritonavir. Also, to assess in a preliminary manner the pharmacokinetics and toxicity profile of BAY 43-9006 in patients who are not receiving ritonavir.

ELIGIBILITY: Key eligibility criteria are as follows: patients 18 years of age or older, with or without HIV infection, and with KS and at least 5 cutaneous lesions untreated by local therapy; patients with HIV infection must have KS that is progressing or stable on highly active antiretroviral therapy (HAART); patients with extensive active, visceral, or symptomatic KS are excluded.

DESIGN: Patients with AIDS-KS who are receiving ritonavir will be administered BAY 43-9006. An initial group of patients will be administered 200 mg BAY 43-9006 once daily, and subsequent groups will receive 200 mg twice daily and 400 mg twice daily respectively. Also two groups of patients with KS and not on ritonavir will be administered 200 mg and 400 mg BAY 43-9006 twice daily respectively. Patients will be studied for toxicity, pharmacokinetics, KS response, the effect on biological markers such as target receptor kinase phosphorylation and signaling molecules in KS tissue. Other parameters that will be assessed will include VEGF levels, the viral load of KSHV, and KS lesion blood flow by non-invasive techniques. If patients tolerate BAY 43-9006, they will receive it for up to 24 weeks. If they have evidence of stable KS or a tumor response, they may receive the drug for up to 54 weeks total.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 years or greater.
  2. Kaposi's sarcoma (KS) pathologically confirmed by CCR Pathology. Patients with both HIV-associated and HIV-negative KS will be eligible.
  3. Either (1) at least 5 measurable cutaneous KS lesions with no previous local therapy, or (2) other measurable non-cutaneous disease that permits a response to be assessed.
  4. Patients with HIV-related KS must be receiving and be willing to comply with a regimen of highly active antiretroviral therapy (HAART) consistent with DHHS treatment guidelines that either (1) utilizes 3 or more drugs or (2) attains suppression of HIV below the limit of detection (50 copies HIV/ml using Roche Amplicor Monitor assay or similar standard test).
  5. For patients with HIV-associated KS, KS lesions must either (1) be increasing during the 3 months prior to screening while the patient is receiving HAART or has unchanged suppression of HIV to below the limits of detection; or (2) must be stable for at least four months while the patient is taking highly active antiretroviral therapy (HAART).
  6. ECOG performance status less than or equal to 2
  7. Life expectancy greater than 6 months
  8. The following hematologic parameters:
* Hemoglobin greater than 9 g/l
* WBC greater than 1000/mm(3)
* Platelets greater than 75,000/mm(3)
* PT and PTT less than or equal to 120% of control, unless the patient has the presence of a lupus anticoagulant

The following hepatic parameters:

* For patients not receiving protease inhibitor therapy: bilirubin less than or equal to 1.5 times the upper limit of normal (ULN). For patients receiving protease inhibitor therapy and for whom the elevated bilirubin is felt to be related to this therapy total bilirubin should be less than or equal to 3.7 mg/dl with a direct fraction less than or equal to 0.2 mg/dl.
* AST/GOT less than or equal to 2.5 times the ULN
* Either serum creatinine less than or equal to 1.5 mg/dl or measured creatinine clearance greater than 60 mL/min.
* Patients must be willing to use effective birth control.

EXCLUSION CRITERIA:

1. Patients with extensive active or symptomatic pulmonary KS
2. Patients with symptomatic visceral KS, except for that involving the oral cavity
3. KS that appears to be improving after other therapy
4. Inability to provide informed consent
5. Patients requiring systemic therapy with ketoconazole or itraconazole
6. Cytotoxic chemotherapy or other specific KS therapy (except for antiretroviral therapy) within the past 3 weeks.
7. Prior therapy with BAY 43-9006
8. Known hypersensitivity to BAY 43-9006
9. Supraphysiologic doses of corticosteroids within 3 weeks
10. Pregnancy (because of unknown potential for fetal malformation)
11. Breast feeding (because of unknown potential for adverse infant developmental considerations)
12. Past or present history of malignant tumors other than KS unless: a) in complete remission for greater than or equal to 1 year from the time a response was first documented; b) completely resected basal cell carcinoma; or c) in situ squamous cell carcinoma of the cervix or anus
13. Evidence of severe or life-threatening infection within 2 weeks of entry into the study
14. Elevated lipase greater than 2 times the ULN or amylase greater than 2 times the ULN (unless documented to be of non-pancreatic origin or associated with macroamylasemia
15. Patients with any other abnormality that would be scored as a grade 3 or greater toxicity, except:

    * lymphopenia
    * direct manifestation of KS
    * direct manifestation of HIV infection, except for neurologic or cardiac manifestations.
    * direct manifestation of HIV therapy, except for neurologic or cardiac manifestations or those addressed elsewhere in the eligibility requirements or that would be scored as grade 4.
    * asymptomatic hyperuricemia
16. Any condition that, in the opinion of the principal Investigator or Study Chairperson would preclude the inclusion of a patient into this research study.
17. Patients must not have evidence of a bleeding diathesis.
18. Patients must not be on therapeutic coagulation. Prophylactic anticoagulation (i.e. low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for PT and PTT are met.
19. Patients must not be taking cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine, and Phenobarbital), rifampin, or St. Johns Wort.
20. Patients are excluded if they have uncontrolled hypertension (diastolic blood pressure greater than 99 mm Hg or systolic blood pressure greater than 159 mm Hg)
21. Patients are excluded if they have uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
22. Patients must be able to understand and be willing to sign a written informed consent document, and express willingness and the ability to comply with the requirements of the protocol.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-02-02; Primary Completion 2012-09-21 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Assess toxicity profile and pharmacokinetics of BAY 43-9006 | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gao SJ, Kingsley L, Li M, Zheng W, Parravicini C, Ziegler J, Newton R, Rinaldo CR, Saah A, Phair J, Detels R, Chang Y, Moore PS. KSHV antibodies among Americans, Italians and Ugandans with and without Kaposi's sarcoma. Nat Med. 1996 Aug;2(8):925-8. doi: 10.1038/nm0896-925. PMID 8705864
- [Background] Biggar RJ, Rosenberg PS, Cote T. Kaposi's sarcoma and non-Hodgkin's lymphoma following the diagnosis of AIDS. Multistate AIDS/Cancer Match Study Group. Int J Cancer. 1996 Dec 11;68(6):754-8. doi: 10.1002/(SICI)1097-0215(19961211)68:63.0.CO;2-0. PMID 8980179
- [Background] Antman K, Chang Y. Kaposi's sarcoma. N Engl J Med. 2000 Apr 6;342(14):1027-38. doi: 10.1056/NEJM200004063421407. No abstract available. PMID 10749966
- [Derived] Uldrick TS, Goncalves PH, Wyvill KM, Peer CJ, Bernstein W, Aleman K, Polizzotto MN, Venzon D, Steinberg SM, Marshall V, Whitby D, Little RF, Wright JJ, Rudek MA, Figg WD, Yarchoan R. A Phase Ib Study of Sorafenib (BAY 43-9006) in Patients with Kaposi Sarcoma. Oncologist. 2017 May;22(5):505-e49. doi: 10.1634/theoncologist.2016-0486. Epub 2017 Mar 24. PMID 28341759